CLINICAL TRIAL: NCT05251155
Title: Accuracy of Mobile-Based Vision Charts in Clinical Practice.
Brief Title: Accuracy of Mobile-Based Vision Charts.
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Other Study IDs: RC-15-2-01
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Visual Spatial Processing
Keywords: Visual acuity; Mobile-based chart; Snellen's chart
MeSH Terms: conditions — Spatial Processing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard vision chart.: Best corrected visual acuity measured by standard chart projector.
  Interventions: Diagnostic Test: Distant best corrected visual acuity assessment
- Mobile based vision chart.: Best corrected visual acuity measured by mobile based chart with screen mirroring over 24 inch monitor.
  Interventions: Diagnostic Test: Distant best corrected visual acuity assessment

INTERVENTIONS:
Diagnostic Test: Distant best corrected visual acuity assessment — Measuring distant visual acuity on snellen's chart using two methods and results were converted to equivalent logarithm of minimum angle of resolution to compare accuracy of mobile based chart to the standard vision chart.

SUMMARY:
Analyzing the accuracy of mobile-based distant vision charts in clinical practice as an economic alternative for standard vision charts.

DETAILED DESCRIPTION:
Accuracy of mobile-based visual acuity testing in clinical practice is still debatable. The aim of this study was to analyze the accuracy of mobile-based distant vision chart in comparison to standard chart projector.

ELIGIBILITY:
Inclusion Criteria:

* Subjects visited ophthalmology clinic at Al-Nil Hospital, Banha, EGYPT for visual acuity assessment.
* Subjects that their best corrected visual acuity was ranged from 0.1 to 1.0 in decimal form measured on snellen's chart.

Exclusion Criteria:

* Subjects that refuse to measure visual acuity twice during the same visit.
* Subjects that their best corrected visual acuity is less than 0.1 in decimal form by the standard chart projector.

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects aimed to asses their best corrected visual acuity or seek spectacles prescription at ophthalmology clinic at Al-Nil Hospital, Banha, EGYPT.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Accuracy of mobile based "snellen chart" in measuring distant visual acuity. | Immediately after visual acuity testing using the standard chart projector.
  To compare the decimal results of mobile based snellen chart for measuring distant vision with the decimal results of the standard snellen chart projector.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Study Chair — Benha University
Locations (1):
- Al-Nil Hospital, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: Undecided